CLINICAL TRIAL: NCT03053167
Title: Irinotecan Plus Raltitrexed as Second-line Treatment in Advanced Colorectal Cancer Patients: An Open-label, Single-arm, Multicenter Phase II Study
Brief Title: Irinotecan Plus Raltitrexed as Second-line Treatment in Advanced Colorectal Cancer Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Collaborators: The First Affiliated Hospital of Dalian Medical University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Shengjing Hospital (Other); General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Director of Department of Medical Oncology，The First Hospital of China Medical University, China Medical University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOG1602
Record Dates: First submitted 2017-01-23; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: ColoRectal Cancer
Keywords: Raltitrexed; Irinotecan; Second-line Treatment; Advanced Colorectal Cancer(ACC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; raltitrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Irinotecan & Raltitrexed (Experimental): advanced colorectal cancer patients treated with irinotecan plus raltitrexed as second-line treatment.
  Irinotecan:180mg/㎡+NS250ml, ivgtt, 90min, d1
  Raltitrexed: 3mg/㎡+NS100ml，ivgtt，15min, d1 Every 3 weeks
  Interventions: Drug: Irinotecan; Drug: Raltitrexed

INTERVENTIONS:
Drug: Irinotecan — Irinotecan: 180mg/㎡+NS250ml, ivgtt, 90min, d1 Every 3 weeks
  Other Names: Campto
Drug: Raltitrexed — Raltitrexed: 3mg/㎡+NS100ml，ivgtt，15min, d1 Every 3 weeks
  Other Names: Sai wei jian

SUMMARY:
Irinotecan and raltitrexed are active against advanced colorectal cancer (ACC), act through different mechanisms, and have only partially overlapping toxicity profiles. The purpose of this study is to evaluate efficacy and safety of irinotecan plus raltitrexed as second-line treatment in advanced colorectal cancer patients.

DETAILED DESCRIPTION:
The standard initial treatment for patients with advanced colorectal cancer (ACC) not amenable for surgical resection is palliative 5-fluorouracil (5-FU)-based chemotherapy. However, response rates are low and prognosis remains poor, with median survival times about one year. Until recently, second-line therapy options were limited.

Irinotecan is a semisynthetic camptothecin derivate that acts as a DNA-topoisomerase-1 inhibitor,its most frequent toxic effects are diarrhea, neutropenia and cholinergic syndrome. Raltitrexed is a quinazoline folate-based specific thymidylate synthase inhibitor, its clinical activity in this setting is similar to that of modulated 5-FU regimens but with a better toxicity profile (mainly asthenia and increased serum transaminase levels). There seems to be no cross-resistance between 5-FU and raltitrexed. Irinotecan and raltitrexed have different toxicity profiles and modes of action. Both drugs are active as single agents and may be given as a short 3-weekly infusion, thus obviating complex schedules or the need for implantable venous access devices. Preclinical studies have demonstrated a pronounced sequence-dependent synergy between SN-38 (the active metabolite of irinotecan) and raltitrexed. It seems then interesting to explore the feasibility and therapeutic potential of this association.

With this background, the investigators have performed this study to evaluate efficacy and safety of irinotecan plus raltitrexed as second-line treatment in advanced colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* life expectancy of at least 3 months;
* histological and/or cytological confirmation of ACC;
* disease progression while on first-line palliative oxaliplatin & fluoropyrimidine chemotherapy or relapse within 6 months after adjuvant oxaliplatin & fluoropyrimidine chemotherapy;
* wash-out time of 4 weeks after the last chemotherapy infusion or radiotherapy，and observed lesions not in the radiotherapy target；
* at least one measurable objective tumor lesion by spiral CT examination, the maximum diameter ≥ 1cm（according to RECIST 1.1）；
* ECOG performance status 0-1；
* satisfactory main organ function，laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count（ANC） ≥1.5×109/L, platelet count（PLT） ≥90×109/L, Serum creatinine（CR）≤1.5 upper normal limitation (UNL)，creatinine clearance rate (CCr) ≥60ml/min, total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL);
* For women with child bearing potential, a negative serum or urine pregnancy test result should be obtained before enrollment
* written informed consent.

Exclusion Criteria:

* prior exposure to irinotecan or raltitrexed;
* chronic enteropathy on unresolved bowel obstruction;
* Pregnant or lactated women;
* previous malignant disease other than carcinoma in situ of the cervix or basal cell carcinoma of the skin;
* Concurrent administration of any other investigational drug, or have been enrolled in other clinical trial with investigational drug treatment within the 30 days of start of study treatment；
* cerebral metastases or leptomeningeal carcinomatosis;
* severe or uncompensated concomitant medical conditions.
* Unsuitable for the study or other chemotherapy determined by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival [PFS] | 5-6 months

SECONDARY OUTCOMES:
Overall Survival [OS] | 12-15 months
Objective Response Rate [ORR] | 12-15 months
Disease Control Rate [DCR] | 12-15 months

OTHER OUTCOMES:
Incidence and Degree of Treatment-Emergent Adverse Events [Safety and Tolerability] | 12-15 months
Performance Status [WHO-ECOG] | 12-15 months
Quality of Life [WHO-QOL] | 12-15 months

CONTACTS AND LOCATIONS:
Overall Officials: YunPeng Liu, PhD, Principal Investigator — First Hospital of China Medical University
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China

REFERENCES:
- [Result] Chiara S, Nobile MT, Tomasello L, Acquati M, Taveggia P, Murolo C, Percivale P, Rosso R. Phase II trial of irinotecan and raltitrexed in chemotherapy-naive advanced colorectal cancer. Anticancer Res. 2005 Mar-Apr;25(2B):1391-6. PMID 15865096
- [Result] Feliu J, Salud A, Escudero P, Lopez-Gomez L, Pericay C, Castanon C, de Tejada MR, Rodriguez-Garcia JM, Martinez MP, Martin MS, Sanchez JJ, Baron MG; Oncopaz Cooperative Group and Associated Hospitals. Irinotecan plus raltitrexed as first-line treatment in advanced colorectal cancer: a phase II study. Br J Cancer. 2004 Apr 19;90(8):1502-7. doi: 10.1038/sj.bjc.6601713. PMID 15083176
- [Result] Aparicio J, de las Penas R, Vicent JM, Garcera S, Llorca C, Maestu I, Yuste AL, Farres J. Multicenter phase I study of irinotecan plus raltitrexed in patients with 5-fluorouracil-refractory advanced colorectal cancer. Oncology. 2002;63(1):42-7. doi: 10.1159/000065719. PMID 12187070
- [Result] Carnaghi C, Rimassa L, Garassino I, Zucali PA, Masci G, Fallini M, Morenghi E, Santoro A. Irinotecan and raltitrexed: an active combination in advanced colorectal cancer. Ann Oncol. 2002 Sep;13(9):1424-9. doi: 10.1093/annonc/mdf229. PMID 12196368
- [Derived] Cheng Y, Teng Z, Zhang Y, Jin B, Zheng Z, Man L, Wang Z, Teng Y, Yu P, Shi J, Luo Y, Wang Y, Zhang J, Zhang H, Liu J, Chen H, Xiao J, Zhao L, Zhang L, Jiang Y, Chen Y, Zhang J, Wang C, Liu S, Qu J, Qu X, Liu Y. Irinotecan plus raltitrexed as second-line treatment in locally advanced or metastatic colorectal cancer patients: a prospective open-label, single-arm, multi-center, phase II study. BMC Cancer. 2024 Sep 2;24(1):1082. doi: 10.1186/s12885-024-12831-4. PMID 39223545